CLINICAL TRIAL: NCT05197738
Title: Research Framework Exploring Sleep Health
Acronym: REFRESH
Status: Recruiting | Type: Observational
Sponsor: Scripps Translational Science Institute (Other)
Responsible Party: Principal Investigator, Stuti Jaiswal, Assistant Professor of Molecular Medicine, Scripps Translational Science Institute
Other Study IDs: IRB-21-7863
Record Dates: First submitted 2021-12-16; First posted 2022-01-19 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Sleep; Sleep Apnea; Obesity; Mood
MeSH Terms: conditions — Sleep Apnea Syndromes; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — An eventual goal of this study is to include a genetic assessment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (11):
- High risk OSA: Cohort of individuals found to sleep have scores categorized as "High risk," on the Berlin questionnaire.
- Low risk OSA: Cohort of individuals found to sleep have scores categorized as "Low risk," on the Berlin questionnaire.
- Short sleepers: Cohort of individuals found to have average sleep duration of < 7 hours per night. Individuals who sleep on average less than 6 hours per night will further be sub-categorized as very short sleeprs.
- Long sleepers: Cohort of individuals found to have average sleep duration of >9 hours per night.
- Average lengths leepers: Cohort of individuals found to have an average sleep duration between 7 and 9 hours per night
- Regular sleepers: Cohort of individuals whose standard deviation of sleep duration falls within 1 standard deviation of their mean sleep duration.
- Irregular sleepers: Cohort of individuals whose standard deviation of sleep duration falls greater than 1 standard deviation of their mean sleep duration
- Severe insomnia risk: Cohort of individuals whose scores on the Insomnia Severity Index would be categorized as severe
- Moderate insomnia risk: Cohort of individuals whose scores on the Insomnia Severity Index would be categorized as moderate
- No insomnia risk: Cohort of individuals whose scores on the Insomnia Severity Index would be categorized as low
- Increased social jet lag: Individuals who are more than 1 hour less or more of sleep on weekdays compared to average weekend sleep.

SUMMARY:
This is a digital health study in which participants are recruited to collect sleep and activity data from digital activity trackers. We are also collecting survey/questionnaire data on baseline health and sleep characteristics as well as bi-weekly assessments of sleep quality and mood. Overall, we aim to examine how sleep relates to physical and mental health in a large population of activity tracker users.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Residing within the United States
* Ability to use the REFRESH app on the participant's own smartphone device

Exclusion Criteria:

* In-ability to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: General adult population.
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2041-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire 9 | Administered one time at enrollment
  Baseline depression scores on a scale from 0 to 27, which higher scores indicated more depression
Bi-weekly mood scores | Averaged bi-weekly over a two month period
  Mood scores based on an 11 point rating scale, with higher scores indicated a better mood
Subjective sleep quality | Averaged bi-weekly over a two month period
  Biweekly assessment of refreshing sleep quality on an 11 point rating scale, with higher scores indicated better subjective sleep from the participant
Change in BMI | Measured as the difference between BMI reported at the beginning of the study and at the two-month mark.
  Based on standard BMI categories; calculated based on self-reported data of height and weight

CONTACTS AND LOCATIONS:
Overall Officials: Stuti Jaiswal, MD, PhD, Principal Investigator — Scripps Research Institute
Locations (1):
- Scripps Research Institute, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Undecided